CLINICAL TRIAL: NCT04341753
Title: Intra- and Inter-evaluator Reproducibility of Upper Limb Strength Measures With Handheld Dynamometer, in Patients With COPD
Brief Title: Intra- and Inter-evaluator Reproducibility of Upper Limb Strength Measures in Patients With COPD
Acronym: FORMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC19.0237
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): In addition to the usual evaluation, other tests will be carried out in addition and specifically for this study:
  * the strength' measure of the deltoids, triceps and brachial biceps will be carried out by another technique: the 1-RM technique (with dumbbells);
  * 2 other times, the strength' measure of the deltoids, triceps and brachial biceps will be carried out by handheld dynaometry.
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — the strength' measure of the deltoids, triceps and brachial biceps will be carried out by another technique: the 1-RM technique (with dumbbells);
  - 2 other times, the strength' measure of the deltoids, triceps and brachial biceps will be carried out by handheld dynaometry.

SUMMARY:
According to the recommendations of French and international learned societies, respiratory rehabilitation is part of the care of patients with Chronic Obstructive Pulmonary Disease (COPD). Indeed, scientific work carried out for more than 10 years on the respiratory rehabilitation of patients suffering from COPD shows that respiratory rehabilitation allows a reduction of the handicap caused by the disease and an improvement in the quality of life of the patients.

A respiratory rehabilitation program (PRR) includes: individual exercise re-training, therapeutic education, respiratory physiotherapy, help with smoking cessation and nutritional and psychosocial care. Exercise retraining includes training the muscles of the lower limbs in endurance and strength combined with training the muscles of the upper limbs. Strengthening the upper limbs helps reduce dyspnea in patients with COPD. In order to determine a precise muscle building protocol, it is necessary to assess at the start of the program the maximum voluntary strength (FMV) of the different muscle groups of the upper limbs. Measuring FMV quantifies a possible frequent strength deficit in patients with COPD and the effects of the strengthening program. Currently, tests to assess FMV using isokinetic dynamometers are used as a benchmark. However, this material is little used in current practice. Portable dynamometers are used to perform simple tests and to obtain muscle strength measurements. However, the reliability of the maximum voluntary force measurements of the different muscle groups of the upper limb has not been evaluated. Studies seem necessary to determine the reproducibility of the measurement in intra and inter-examiner (Schrama 2014) and to assess its sensitivity to change during a respiratory rehabilitation program. The objectives of this study are to study the reproducibility, validity and sensitivity to change of the measurement of FMV using a portable dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD stages 2 to 4 (A to D) admitted to the pulmonary rehabilitation unit of Centre Hospitalier des Pays de Morlaix (4 weeks)
* Patient able to consent and having signed a consent form
* Patient 18 years of age or older

Exclusion Criteria:

* Patient with pain, arthritis, prosthetics, shoulder or elbow surgery.
* Patient with a history of pneumonectomy, lobectomy less than 6 months old
* Refusal to participate
* Patient with an inability to follow a full respiratory rehabilitation program
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Change isometric voluntary muscle strength measure, with hand held dynamometer | up to 4 weeks
  the strength of the deltoid, biceps, triceps muscles is measured with handheld dynamometer, 3 times

SECONDARY OUTCOMES:
isometric voluntary muscle strength measure, with the one repetition of maximal resistance (1-MR) test (with dumbbells) | up to 4 weeks
  the strength of the deltoid, biceps, triceps muscles is measured with 1-MR test
isometric voluntary muscle strength measure, with hand held dynamometer | 4 weeks
  the strength of the deltoid, biceps, triceps muscles is measured with handheld dynamometer, a te the beginning and and the end of the pulmonary rehabilitation program
the 6-minute walk test | up to 4 weeks
  The improvement in exercise capacity is measured in the 6-minute walk test
1-minute sit to stand test | up to 4 weeks
  The improvement in exercise capacity is measured during a 1-minute sit to stand test
The voluntary force of the quadriceps | up to 4 weeks
  the maximum voluntary force of the quadriceps is measured with a MICROFET dynamometer
he endurance time of quadriceps | up to 4 weeks
  the improvement of the endurance time of quadriceps is mesured with a MICROFET dynamometer
The dyspnea sensation by Modified Medical Research Council scale | up to 4 weeks
  The improvement in dyspnea sensation is measured with the Modified Medical Research Council scale This unidimensional scale is used to assess dyspnea in the daily life of a patient from stage 0 to stage 4.
The dyspnea sensation by LCADL questionnaire | up to 4 weeks
  he improvement in dyspnea sensation is measured with the LCADL questionnaire The purpose of this questionnaire is to help understand how the patient perceives and feels your breathing with a score from 0 to 75
the dyspnea sensation by dypsnea-12 scale | up to 4 weeks
  The improvement in dyspnea sensation is measured with the dypsnea-12 scale. This questionnaire is used to evaluate the physical and emotional aspects of dyspnea with 12 questions.
the dyspnea sensation by MDP questionnaire | up to 4 weeks
  The improvement in dyspnea sensation is measured with the MDP questionnaire This questionnaire makes it possible to measure the discomfort, the sensory qualities of the dyspnea, the intensity of the sensations, the emotional sensations.
Quality of life by CAT questionnaire | up to 4 weeks
  The improvement in quality of life is measured with CAT questionnaire. The CAT is one component in clinical decision-making, along with other considerations such as history of previous exacerbations and airflow limitation. A score is calculated from 8 questions with an answer from 0 to 5.
Quality of life by St Georges questionnaire | up to 4 weeks
  The improvement in quality of life is measured with St Georges questionnaire This questionnaire is a self-reported disease-specific, health-related quality of life questionnaire. It was originally developed to measure the impact of Chronic Obstructive Pulmonary Disease on a person's life, but has also been studied and applied to non-COPD pulmonary populations.
Fear of falling | up to 4 weeks
  The decrease in fear of falling is measured with the FES-I questionnaire. This questionnaire evaluates the fear of falling with a score from 0 to 30.
Anxiety and depression | up to 4 weeks
  The evolution of anxiety and depression is measured with HAD scale This scale is an instrument for screening for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions are related to the anxiety dimension (total A) and seven others to the depressive dimension (total D), allowing two scores to be obtained (maximum score of each score = 21).
Self-esteem | up to 4 weeks
  The changes in self-esteem are measured with ISP-6 questionnaire This questionnaire is a 6-question questionnaire on overall self-esteem giving a score of
Evolution of the non fat mass index | up to 4 weeks
  The evolution of the non fat mass index is measured with impedancemetry

CONTACTS AND LOCATIONS:
Overall Officials: Loïc PERAN, Principal Investigator — CH des pays de Morlaix
Locations (1):
- Centre Hospitalier des pays de Morlaix, Morlaix, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH will be required to sign and complete a data access agreement

REFERENCES:
- [Background] Awatani T, Morikita I, Shinohara J, Mori S, Nariai M, Tatsumi Y, Nagata A, Koshiba H. Intra- and inter-rater reliability of isometric shoulder extensor and internal rotator strength measurements performed using a hand-held dynamometer. J Phys Ther Sci. 2016 Nov;28(11):3054-3059. doi: 10.1589/jpts.28.3054. Epub 2016 Nov 29. PMID 27942118
- [Background] Nyberg A, Saey D, Maltais F. Why and How Limb Muscle Mass and Function Should Be Measured in Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2015 Sep;12(9):1269-77. doi: 10.1513/AnnalsATS.201505-278PS. PMID 26208090
- [Derived] Peran L, Berriet AC, Le Ber C, Consigny M, Beaumont M. Reliability and Validity of Upper Limb Muscle Strength Measurements by Handheld Dynamometer in Patients With Chronic Obstructive Pulmonary Disease. Physiother Res Int. 2025 Oct;30(4):e70111. doi: 10.1002/pri.70111. PMID 40991671